CLINICAL TRIAL: NCT02970084
Title: Role of Vitamin K2 in the Reduction of the Calcium Content at the Level of the Carotid Bifurcation in Patients With Subcritical Lesions
Brief Title: Vitamin K2 for Reduction the Calcium at Carotid Bifurcation in Patients With Subcritical Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, yamume tshomba, Medical doctor Associate Professor of Vascular Surgery, Scientific Institute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PLAK2/74/OSR
Record Dates: First submitted 2016-11-18; First posted 2016-11-21 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Carotid Plaques

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Group with K2 (Experimental): The nutraceutical product (PLAK2) based on vitamin K2, will be administered once a day (a tablet 800mg) for 12 months.
  All patients enrolled will continue to be treated according to the clinical standard (100 mg Cardioaspirin, cp 1 day : Acetylsalicylic acid)
  Interventions: Other: Nutraceutical product based on vitamin K2 (PLAK2)
- Control group (no vitamin K2) (No Intervention): The control group did not take the supplement of Vitamin K2. All patients enrolled will continue to be treated according to the clinical standard (100 mg Cardioaspirin, cp 1 day : Acetylsalicylic acid)

INTERVENTIONS:
Other: Nutraceutical product based on vitamin K2 (PLAK2)
  Other Names: PLAK2
  Arms: Group with K2

SUMMARY:
Clinical study single center, prospective, randomized, controlled (vs. no supplement), open-label, blinded assessor (the doctor who will perform the Doppler ultrasound at 6 and 12 months will not know the treatment given to the patient, because the diagnostic test in question is considered operator-dependent), a "parallel group", which aims is evaluate the reduction in the level of calcium in the carotid artery and the carotid atherosclerotic plaques, on a sample of 60 subjects presenting subcritical calcified lesions of the carotid bifurcation with a range of 40-60%.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Ability to provide written informed consent
3. subjects with calcified lesions subcritical from the carotid bifurcation. with a range of 40-60% calculated method with ECTS (European Carotid Surgery Trial)

Exclusion Criteria:

1. Patients with reduced life expectancy or age> 80 years,
2. Patients already subjected to other clinical trial in the previous three months,
3. Patients with hypersensitivity or with known allergies to acetylsalicylic acid, patients with pre-existing mastocytosis, a history of asthma induced by salicylates, duodenal ulcer, bleeding diathesis, severe hepatic insufficiency, severe heart failure, concomitant treatment with methotrexate, last trimester of pregnancy.
4. Patients with known hypersensitivity to vitamin K2 and vitamin D, people with hemolytic diseases, concomitant anticoagulant therapy, people with cancer, MAV (arteriovenous malformations) and / or cerebral aneurysms, hypercalcemia, nephrolithiasis and renal failure.
5. Uncooperative patients , or allergies related to the substance under study or with any contra-indicated in the data sheet / Summary of Product Characteristics (SPC) of the substances in the studio.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Reduction of calcium content, to 12 months, at the level of carotid atheromatous plaque | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Italy